CLINICAL TRIAL: NCT04676997
Title: A Phase Ⅱ Study to Evaluate Efficacy and Safety of Camrelizumab Plus Chemotherapy as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC)
Brief Title: Neoadjuvant Study of Camrelizumab Plus Chemotherapy in Triple Negative Breast Cancer (TNBC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinming Yu, Director of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-006
Record Dates: First submitted 2020-11-30; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: Neoadjuvant; PD-1
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; Taxes; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Chemotherapy (Experimental): Participants receive Camrelizumab d1,15 (Q2W) + nab-paclitaxel d1,8,15(QW 3/4) x 4 cycles, followed by Camrelizumab Q2W + epirubicin + cyclophosphamide Q2W x 4 cycles as neoadjuvant therapy prior to surgery
  Interventions: Biological: Camrelizumab; Drug: Nab paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Camrelizumab — 200mg on days1,15 of Cycles 1-4 (Q2W); IV infusion. 200mg on day 1 of Cycles 5-8 (Q2W); IV infusion.
Drug: Nab paclitaxel — 125 mg/m² on day 1, 8 and 15 of Cycles 1-4 (QW 3/4); IV infusion.
Drug: Epirubicin — 90 mg/m² on day 1 of Cycles 5-8 (Q2W); IV infusion.
Drug: Cyclophosphamide — 600 mg/m² on day 1 of Cycles 5-8 (Q2W); IV infusion.

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of Camrelizumab Combination With Nab-Paclitaxel and Epirubicin as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC)

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed breast cancer
2. 18-70 Years, female;
3. life expectancy is not less than 3 months
4. Histologically documented TNBC (negative human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PgR] status);
5. Stage at presentation: T1c N1-2 or T2-4 N0-2;
6. at least one measurable lesion according to RECIST 1.1;
7. Adequate function of major organs meets the following requirements:

   * Neutrophils ≥ 1.5×10^9/L
   * Platelets ≥ 100×10^9/L
   * Hemoglobin ≥ 90g/L
   * lymphocyte≥0.5×10^9/L
   * Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
   * ALT and AST ≤ 3 × ULN
   * ALP≤ 2.5 × ULN
   * BUN and Cr ≤ 1.5 × ULN
   * TSH≤ ULN
   * Left ventricular ejection fraction (LVEF) ≥ 50%
   * QTcF ≤ 470 ms
8. Provides tumor tissue specimen to assess tumor programmed death-ligand 1 (PD-L1);
9. For women of childbearing potential: agreement to use contraceptive methods. Women who are not postmenopausal or have undergone a sterilization procedure must have a negative serum pregnancy test result within 72 hours prior to initiation of study drug.

Exclusion Criteria:

1. Stage Ⅳ (metastatic) breast cancer or bilateral breast cancer
2. Inflammatory breast cancer
3. patients who received chemotherapy, endocrine therapy, immunotherapy, biotherapy or TACE within 4 weeks before admission
4. Has participated in an interventional clinical study with an investigational compound within 4 weeks prior to initiation of study treatment
5. Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies
6. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
7. Major surgical procedure within 4 weeks prior to initiation of study treatment
8. Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus
9. Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases
10. Administration of a live attenuated vaccine within 28 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study
11. Has a known history of Human Immunodeficiency Virus (HIV).
12. Has known active Hepatitis B, Hepatitis C or Autoimmune hepatitis
13. Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
14. Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment
15. Has evidence of active tuberculosis within 1year prior to initiation of study treatment
16. Prior allogeneic stem cell or solid organ transplantation
17. Pre-existing motor or sensory neuropathy of a severity≥grade 2
18. Has significant cardiovascular disease
19. Treatment with systemic immunostimulatory agents within 4 weeks prior to initiation of study treatment
20. Treatment with systemic immunosuppressive medications within 2 weeks prior to initiation of study treatment
21. Has a known hypersensitivity to the components of the study treatment or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
22. Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial
23. History of neurological or psychiatric disorders, including epilepsy or dementia.
24. any other situation evaluated by researchers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
pCR rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive tumor on hematoxylin and eosin evaluation of breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.

SECONDARY OUTCOMES:
pCR rate using the definition of ypT0/Tis (i.e., absence of invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants
Event-Free Survival (EFS) in all participants | Up to approximately 5 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Objective Overall Response Rate (ORR) | Up to approximately 25-30 weeks
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until definitive surgery or disease progression.
Adverse events (AEs) | Up to approximately 35 weeks
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Center, Shandong Cancer Hospital Affiliated to Shandong University Recruiting, Jinan, Shandong, China